CLINICAL TRIAL: NCT03819348
Title: The First Affiliated Hospital of Guangxi Medical University
Brief Title: Retrospective Analysis of the Epidemiological Change and Determinants of Prognosis of Talaromycosisof Human Immunodeficiency Virus Negative Host in Guangxi
Acronym: RAECDPT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Guangxi Medical University (Other)
Collaborators: Second Affiliated Hospital of Guangzhou Medical University (Other); The Fourth People's Hospital of Nanning (Other); Guilin Medical College (Other); Nanning Second People's Hospital (Other); People's Hospital of Guangxi Zhuang Autonomous Region (Other)
Responsible Party: Principal Investigator, Qiu Ye, Professor, Guangxi Medical University
Other Study IDs: RA-TSM-HIVN-ECDP
Record Dates: First submitted 2019-01-15; First posted 2019-01-28 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: To Investigate the Characteristics and Prognostic Factors of T. Marneffei Infections and the Causes of Misdiagnosis; To Study the Recurrence Indicators and Establish a Therapeutic Effect Evaluation System of T. Marneffei Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TSM of HIV-negative Host: Eligible patients were HIV-infected adults who had talaromycosis that was confirmed by either microscopy or culture.
  Interventions: Other: the multiple programs of antifungal therapy for HIV-negative host

INTERVENTIONS:
Other: the multiple programs of antifungal therapy for HIV-negative host — the multiple programs of antifungal therapy for HIV-negative host TSM were compared in terms of effect on clinical remission rate, effective rate, recurrence rate, mortality and toxic side effects on HIV-negative host TSM; their prognosis and recurrence indicators were clarified, and a therapeutic effect evaluation system was established, providing a standard treatment and diagnosis scheme for clinical practice; and simultaneously the positive rate of G and GM experiments in respect of TSM, Aspergillus and other fungi was identified to provide TSM with biological diagnostic indicators.
  Other Names: their prognosis and recurrence

SUMMARY:
Through a multi-center large-sample retrospective study, the epidemiological changes of TSM in Guangxi have been reviewed, its incidence trend was understood to attract the attention of clinicians; the multiple programs of antifungal therapy for HIV-negative host TSM were compared in terms of effect on clinical remission rate, effective rate, recurrence rate, mortality and toxic side effects on HIV-negative host TSM; their prognosis and recurrence indicators were clarified, and a therapeutic effect evaluation system was established, providing a standard treatment and diagnosis scheme for clinical practice; and simultaneously the positive rate of G and GM experiments in respect of TSM, Aspergillus and other fungi was identified to provide TSM with biological diagnostic indicators. Improve the level of understanding and diagnosis and treatment of HIV-negative TSM in the whole area. A comprehensive efficacy evaluation system and standard treatment program was established to provide a basis for standardized treatment of TSM in HIV-negative hosts. The observational indicators included: 2-week all-cause mortality; 24-week all-cause mortality; clinical improvement time; level of decrease of fungus in the blood culture medium two weeks before treatment; recurrence; appearance of adverse drug reaction at the level 3 and above.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients were HIV-negative adults who had talaromycosis that was confirmed by either microscopy or culture.

Exclusion Criteria:

* patients were HIV-infected adults who had talaromycosis that was confirmed by either microscopy or culture.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We studied the clinical characteristics and prognoses of patients with infections due to Talaromyces marneffei who were admitted to Guangxi Hospital, This province is located in subtropical southern China, where Talaromyces marneffei is endemic.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2003-01-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
clinical remission rate | 7 days
  Clinical resolution of talaromycosis was defined as a temperature of less than 38°C (100°F) for 3 days, resolution of skin lesions, and sterile blood cultures.
recurrence rate | 12 months
  Relapse of talaromycosis was defined as the recurrence of symptoms and a positive fungal culture from any sterile site that led to reinduction of therapy in patients who had achieved clinical resolution.
mortality at 4 week | 4 weeks
  all-cause mortality was defined as the absolute risk of death from any cause during the first 2 weeks after randomization.
toxic side effects | 24 weeks
  Side effects were monitored clinically and with the use of hematologic, chemical, and liver-enzyme testing performed at least twice weekly
mortality at week 24 | 24 weeks
  The secondary outcome measures were mortality at week 24, the time to clinical resolution of talaromycosis, early fungicidal activity, relapse of talaromycosis, and the incidence of adverse events of grade 3 or higher.

SECONDARY OUTCOMES:
G test | 3 days
  positive was defined as >20pg/ml
GM test | 3 days
  positive was defined as >0.5

CONTACTS AND LOCATIONS:
Locations (1):
- Guangxi Medical University, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Le T, Kinh NV, Cuc NTK, Tung NLN, Lam NT, Thuy PTT, Cuong DD, Phuc PTH, Vinh VH, Hanh DTH, Tam VV, Thanh NT, Thuy TP, Hang NT, Long HB, Nhan HT, Wertheim HFL, Merson L, Shikuma C, Day JN, Chau NVV, Farrar J, Thwaites G, Wolbers M; IVAP Investigators. A Trial of Itraconazole or Amphotericin B for HIV-Associated Talaromycosis. N Engl J Med. 2017 Jun 15;376(24):2329-2340. doi: 10.1056/NEJMoa1613306. PMID 28614691
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/28614691